CLINICAL TRIAL: NCT03459118
Title: The Impact of Dementia on Care and Outcomes Associated With a Function Focused Care Intervention Among Residents in Assisted Living Settings.
Brief Title: Dissemination and Implementation of Function Focused Care for Assisted Living
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Barbara Resnick, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 122345; 1R01NR015982-01A1 (NIH)
Record Dates: First submitted 2018-02-24; First posted 2018-03-08 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Dementia; Pain
MeSH Terms: conditions — Dementia; Pain

STUDY DESIGN:
Intervention Model Description: This is an intervention study testing Function Focused Care. The supplement, however, addresses a subsample of the population with dementia and explore the impact of pain on function and behavior and explores if this is a differential impact of the intervention between those with and without dementia. It is a descriptive study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Function Focused Care (Experimental): FFC-AL-EIT is implemented by a Research Nurse Facilitator working with the champion and stakeholders using our four step approach: (I) Environment and Policy Assessments; (II) Education; (III) Establishing Resident Function Focused Care Service Plans; and (IV) Mentoring and Motivating.
  Interventions: Behavioral: Function Focused Care
- Education Only (Placebo Comparator): Education only sites are exposed to Step II of the Four step approach described under the treatment arm. They receive baseline education of staff.
  Interventions: Behavioral: Function Focused Care

INTERVENTIONS:
Behavioral: Function Focused Care — The intervention in the parent study involves the use of a participatory implementation approach as delineated in the Evidence Integration Triangle. Prior to implementation, we meet with the administrator, service coordinator, delegating or oversight nurse or setting contact designee to identify the setting champion and stakeholder team members. In addition to the champion, we recommend the following individuals be included in the stakeholder team: an administrator in a leadership position (e.g. assisted living manager, delegating/overseeing nurse); a direct care worker; a family member; an activity staff member if available; and a resident. FFC-AL-EIT is implemented by a Research Nurse Facilitator working with the stakeholders using our four step approach: (I) Environment and Policy Assessments; (II) Education; (III) Establishing Resident Function Focused Care Service Plans; and (IV) Mentoring and Motivating.

SUMMARY:
This study will evaluate pain, management of pain, behavioral symptoms, and the quality of staff-resident interactions between residents with and without dementia, test the relationship of these variables to participation in function focused care at baseline, and consider if there is a differential impact of FFC-AL-EIT between those with and without dementia with regard to participation in function focused care, functional outcomes and physical activity over the 12 month study period. Findings from this study will provide new information on how to optimize function and physical activity among older adults with dementia in assisted living.

DETAILED DESCRIPTION:
Estimates derived from National data indicate that seven out of ten residents in assisted living have some form of dementia, with 29% having mild impairment, 23% with moderate impairment, and 19% with severe impairment. More than one-third of these residents display behavioral symptoms commonly associated with dementia, approximately 30-50% experience pain, the majority require assistance with activities of daily living (ADLs) and instrumental activities of daily living (IADLs), are sedentary and have limited opportunities to engage in physical activity. Innovative approaches are needed to help residents with dementia remain in assisted living settings. Typically, however, the care of older adults with dementia living in assisted living settings has followed a "just get it done" approach. The focus of care is on task completion and minimization of behavioral symptoms. This results in care that ignores what the resident is able to do for him or herself and is custodial. Residents are not encouraged to perform activities such as combing their own hair, brushing their teeth, or ambulating. Providing custodial care facilitates a decline in physical capability and function, causes medical complications, exacerbates depressive symptoms, increases the likelihood of sustaining a fall and ultimately may result in a need to be transferred to acute or skilled nursing care. To overcome custodial care we use an approach referred to as Function Focused Care. Function Focused Care is a philosophy of care in which staff members engage residents in physical activity at their highest level of ability during all care interactions. Prior research has repeatedly supported the effectiveness of Function Focused Care in terms of maintaining function and increasing time spent in physical activity among older adults in assisted living settings. We do not know, however, if: (1) there is a difference between those with and without dementia in pain, pain management, behavioral and affective symptoms, or the quality of staff-resident interactions; (2) these factors are associated with participation in function focused care activities at baseline; or (3) there is a differential impact of the Function Focused Care for Assisted Living using the Evidence Integration Triangle Intervention (FFC-AL-EIT) between those with and without dementia in terms of participation in function focused care activities, function and physical activity over the 12 month study period. To answer these questions we propose adding measures for pain, behavioral and affective symptoms and quality of staff-resident interactions to Cohort 2 of the parent study, Testing the Dissemination and Implementation of Function Focused Care (1R01AG050516-01A1). The findings from this study will add to what is currently known about older adults with dementia in assisted living and will be used to revise the FFC-AL-EIT intervention as needed to optimize participation in function focused care activities and thereby maintain and improve function and physical activity among older adults with dementia in assisted living.

ELIGIBILITY:
Inclusion Criteria:Residents are eligible to participate if: (1) they are living in a participating assisted living setting and are 65 years of age or older; (2) score at least a one out of three on the three out of three word recall question within the Minicog; and (3) are not enrolled in Hospice.

Exclusion Criteria: Residents will be excluded from the study if they are younger than 65 years of age and do not answer at least one out of three on the three out of three word recall question within the minicog.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 853 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Pain Verbal Descriptor Scale | baseline
  Pain scale that allows respondent to state pain intensity and location
PAINAD | baseline
  an observation measure of pain for individuals with cognitive impairment
Cornell Scale for Depression in Dementia | baseline
  a 19 item survey that assesses depressive symptoms
Resistiveness to Care | baseline
  13 item Likert observation scale of resistiveness to care
Quality of Interaction Scale | baseline
  Observation scale of the positive and negative interactions between staff and residents
Checklist for Evidence of Use of Function Focused Care in the Service Plan | baseline
  Addresses four areas focused on function in the resident's care plan
The Barthel Index | baseline
  A 10-item observation measure of basic activities of daily living
Motionwatch 8 | baseline
  Actigraphy collected for a 5 day period with three full days of data used
Function Focused Care Behavioral Checklist for Residents | baseline
  a 19-item measure that addresses performance by the resident of function focused care

OTHER OUTCOMES:
The Saint Louis University Mental Status Examination (SLUMS) | baseline
  a measure of cognitive ability

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Maryland, Baltimore, Maryland
  - Penn State University, State College, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
will share data based on request and following the development of a IPD sharing plan with the IRB.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At the end of the 5 year study period for the full parent study
Access Criteria: Identification of the purpose for wanting the data

REFERENCES:
- [Derived] McPherson R, Resnick B, Galik E, Gruber-Baldini AL, Holmes S, Kusmaul N. Considerations for Use of the Cornell Scale for Depression in Dementia Among Assisted Living Residents: Factor Analysis Results. J Appl Gerontol. 2025 Dec;44(12):1972-1980. doi: 10.1177/07334648251318783. Epub 2025 Feb 26. PMID 40009165